CLINICAL TRIAL: NCT05729087
Title: Feasibility, Acceptability, and Potential Effectiveness of a Web and Center-based Blended Lifestyle Intervention to Promote Physical Activity, Diet, and Health in Hong Kong Community-dwelling Older Adults: A Pilot Study.
Brief Title: Development of a Blended Lifestyle Intervention to Promote Physical Activity, Diet, and Health in Hong Kong Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Yanping DUAN, Dr. Yanping Duan, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/21-22/0485
Record Dates: First submitted 2022-11-15; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Health Behavior; Physical Activity; Healthy Diet
Keywords: face-to-face intervention; eHealth intervention; health behavior change; old adults
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended Intervention Group (Experimental): A 10-week lifestyle intervention will be provided, addressing physical activity (PA) and healthy diet simultaneously. The program mode is a web- and center-based blended intervention. The web-based lifestyle behavior intervention will be developed based on the Health Action Process Approach.
  Interventions: Behavioral: Blended intervention group
- Control Group (No Intervention): No treatment will be provided during the intervention period. Relevant intervention materials are accessible and available for all participants in the control group after the completion of data collection.

INTERVENTIONS:
Behavioral: Blended intervention group — Face-to-face workshops will be delivered in the neighborhood elderly center every week. Each workshop will consist of two sections (a) a 60-minute PA session, including a Health talk (20 minutes), and a physical exercise training (40 minutes); and (b) a 60-minute healthy diet promotion, including group discussion and sharing (30 minutes), and knowledge of diet and nutrition (30 minutes).
  In addition, a 15-minute online psychological session will be implemented following the PA and diet session.
  Arms: Blended Intervention Group

SUMMARY:
This pilot study will provide a theory-based low-cost and easy-to-operate program in the area of healthy lifestyle promotion among community dwelling older adults. The blended intervention product will be helpful for health professionals, social workers and practitioners working in the elderly centers and health centers to promote older adults' PA, healthy diet and wellness. Furthermore, this study would initiate advocacy for policymakers to disseminate cost-saving, time-efficient and effective healthy lifestyle programs to the communities for healthy aging promotion.

DETAILED DESCRIPTION:
Project Objectives

1. To review and meta-analyze lifestyle interventions for promotion of physical activity, diet and health among older adults.
2. To assess the feasibility of the pilot study.
3. To assess acceptability of the pilot study.
4. To examine between-group differences in changes of physical activity (min/week), diet (portion/day), physical health-related outcomes (physical fitness, blood pressure, fasting blood sugar, and blood lipids), mental health-related outcomes (depression, loneliness) and health-related quality of life (QoL) among the sample.

A series of generalized linear mixed models (GLMM) will be applied to evaluate the intervention effects on outcome measures at T2, with time, groups, and their interaction as fixed effects. Per-protocol analyses will be used for primary analyses, while intention-to-treat approach will be used for sensitivity tests.

ELIGIBILITY:
Inclusion Criteria:

* aged 65-79 years;
* have access to the internet and smartphone;
* speak Cantonese;
* pass the Physical Activity Readiness-Questionnaire (PAR-Q) screening or have the physician's approval prior to participation.

Exclusion Criteria:

* no cognitive disorders or impairments;
* unable to engage in physical activity;

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Change of weekly Physical activity (minutes per week) | Change from baseline to10 week follow-up
  Walking; moderate physical activity; vigorous physical activity The waist-worn accelerometer will be used to objectively assess PA (GT3X+, ActiGraph Inc, Pensacola, FL, USA).
  The Chinese version of the International Physical Activity Questionnaire-short form (IPAQ-C).
  If there is an increase, the result means a better outcome.
Change of Fruit and Vegetable Intake (portions/day) | Change from baseline to10 week follow-up
  To assess the fruit and vegetable intake during the past seven days, participants will be asked "how many portions of fruit they have today" and "how many portions of vegetables they have today". Participants were asked to keep a record for seven days, then to get an average for each day.
  If there is an increase, the result means a better outcome.
Change of Meat, Fish, Egg & Alternatives (MFEA) (taels/day) | Change from baseline to10 week follow-up
  To assess the Meat, Fish, Egg & Alternatives consumption, individuals will be asked to answer three items. To assess the Meat, Fish, Egg & Alternatives during the past seven days, participants will be asked "how many taels of meat do they have today", "how many taels of eggs do they have today" and "how many taels of Alternatives do they have today". Participants were asked to keep a record for seven days, then to get an average intake of Meat, Fish, Egg & Alternatives for each day.
  If there is a change, and the follow-up result is between 5 and 6, the result is better.

SECONDARY OUTCOMES:
Change of Blood pressure (mmHg) | Change from baseline to10 week follow-up
  The Blood pressure will be measured by an automated portable device .
  If there is a change, and the follow-up result is below 120, the result is better.
Change of the Glycosylated Hemoglobin (HbA1c; %) | Change from baseline to10 week follow-up
  The Glycosylated Hemoglobin (HbA1c) will be tested by the Point of Care Cobas b 101 system.
  If there is a change, and the follow-up result is below 6.5, the result is better.
Change of the lipid (mmol/L) | Change from baseline to10 week follow-up
  The lipid, including total cholesterol (CHOL; mmol/L), triglycerides (TG; mmol/L); high-density lipoprotein (HDL; mmol/L); and low-density lipoprotein (LDL; mmol/L)will be tested by Point of Care (POC) Cobas b 101 system.
Change of Agility and dynamic balance | Change from baseline to10 week follow-up
  8 Foot Up-and-Go Test (second)
Change of Upper body flexibility | Change from baseline to10 week follow-up
  Back Scratch Test (upper body; +/- cm)
Change of Lower body flexibility | Change from baseline to10 week follow-up
  Chair Sit and Reach Test (lower body; +/- cm)
Change of Aerobic endurance | Change from baseline to10 week follow-up
  2-Minute Step Test (times in two minutes)
Change of Upper body strength | Change from baseline to10 week follow-up
  30-Second Arm Curl test (upper body; times per 30 seconds)
Change of Lower body strength | Change from baseline to10 week follow-up
  30-Second Chair Stand test (lower body; times per 30 seconds);
Change of Body mass index (kg/m2) | Change from baseline to10 week follow-up
  Body mass index (kg/m2).
Change of Health-Related Quality of life (HRQoL) | Change from baseline to10 week follow-up
  The Hong Kong brief version of the World Health Organization's Quality of Life questionnaire. We measured general quality of life with the question "How would you rate your quality of life?" with a 5-point scale (1=very poor; 5=very good). We also used the physical health subdomain with 7 items, such as "How satisfied are you with your ability to perform your daily living activities?" (1=very dissatisfied; 5=very satisfied).
  If there is an increase, the result means a better outcome.
Change of Depression level (score) | Change from baseline to10 week follow-up
  Geriatric Depression Scale 15-item - Cantonese Version. Participants were asked to indicate the frequency of symptoms on a yes/no questionnaire (yes=1; no=0; except items 1,5,7,9,11: yes=0; no=1) within the last week. Positively formulated items were reversed. The total score consisted of the sum of all 15 items and ranged from 0 to 15. A total score of 5 or greater indicated the likelihood of depression symptoms.
  If there is an increase, the result means a worse outcome.
Change of Loneliness (score) | Change from baseline to10 week follow-up
  The Chinese translation of the 6-item De Jong Gierveld Loneliness Scale. The emotional loneliness was measured by 3 items (yes=1, moderate=1, no=0), such as "I experience a general sense of emptiness". Social loneliness was measured by 3 items (yes=0, moderate=1, no=1). A total score of 2 or greater indicated the likelihood of loneliness.
  If there is an increase, the result means a better outcome.
Change of Self-efficacy of PA and diet | Change from baseline to10 week follow-up
  We assessed self-efficacy for PA with 5 items on a 5-point scale (1=don't agree at all; 5=totally agree), such as "I am certain that I can permanently be physically active for at least 5 days a week for 30 minutes each day".
  We assessed self-efficacy for fruit and vegetable by 5 items on the basis of the PA scale, such as "I am certain that I can eat 5 portions of fruit and vegetables a day even if it is sometimes difficult".
  We assessed self-efficacy for MFEA by 5 items on the basis of the PA scale, such as "I am certain that I can eat moderate MFEA a day even if it is sometimes difficult".
  If there is an increase, the result means a better outcome.
Action control of PA and diet | baseline, 10 week follow-up
  We assessed action control for PA with 6 items on a 5-point scale (1=don't agree at all; 5=totally agree), such as "I consistently monitored when, where, and how long I exercise".
  We assessed action control for FVI/MFEA with 6 items separately on a 5-point scale (1=don't agree at all; 5=totally agree), such as "I consistently monitored whether I ate enough fruit and vegetable /moderate meat".
  If there is an increase, the result means a better outcome.
Change of Planning of PA and diet | Change from baseline to10 week follow-up
  We distinguished planning as action planning and coping planning. We assessed action planning by the stem "For the next month I have carefully planned..." followed by 3 items for PA, such as "which PA I will pursue," and followed by 1 item for FVI and 1 item for MFEA, such as "what I will eat".
  We assessed coping planning by the stem "For the next month I have carefully planned..." followed by 3 items for PA, such as "what I can do in difficult situations to stick to my intentions," or followed by 3 items for FVI and 3 items for MFEA, such as "how I can eat healthy, even if something happened" . Answers were given on a 5-point scale ranging from 1=totally disagree to 5=totally agree.
  If there is an increase, the result means a better outcome.
Change of Social support of PA and diet | Change from baseline to10 week follow-up
  We assessed social support with 3 items for PA and with 3 items for FVI and 3 items for MFEA, such as "My partner helps me/my family helps me/my classmates and friends help me to stay physically active," or "My partner helps me/my family helps me/my classmates and friends help me to eat healthily." Answers were measured with a 5-point scale (1=not at all true; 5=exactly true).
  If there is an increase, the result means a better outcome.
Demographic information | baseline, 10 week follow-up
  Items will include gender, year of birth, marital status, educational level, household income, professional status, living status, number of children, and history of chronic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Duan, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong Baptist University, Kowloon Tong, Hong Kong